CLINICAL TRIAL: NCT00466895
Title: Phase I Study of Lenalidomide in Acute Leukemias and Chronic Lymphocytic Leukemia.
Brief Title: Lenalidomide in Acute Leukemias and Chronic Lymphocytic Leukemia.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Leslie Andritsos (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor-Investigator, Leslie Andritsos, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-06003; NCI-2011-03218 (Other: CTRP (Clinical Trials Reporting Program))
Record Dates: First submitted 2007-04-26; First posted 2007-04-27 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Chronic Lymphocytic Leukemia
Keywords: Leukemia; Lenalidomide
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stratum 1 Acute Leukemias (Experimental): Patients must have a diagnosis of Acute Myeloid Leukemia (AML) or Acute Lymphoblastic Leukemia(ALL)according to the WHO (World Health Organization) classification.
  Interventions: Drug: lenalidomide
- Stratum 2 Chronic lymphocytic leukemia (Experimental): Patients must have diagnosis of B-Cell, Chronic Lymphocytic Leukemia(CLL) or Small Lymphocytic Leukemia (SLL) (including Waldenstrom's Macroglobulinemia) requiring therapy (see eligibility criteria for definition of this) and have previously received treatment with one or more prior chemotherapy regimens.
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — Dose level -1: 2.5 mg daily for days 1-7, 2.5 mg daily for days 8-21. Dose level 1: 2.5 mg daily for days 1-7, 5 mg daily for days 8-21. Dose level 2: 2.5 mg daily for days 1-7, 7.5 mg daily for days 8-21. Dose level 3: 2.5 mg daily for days 1-7, 10 mg daily for days 8-21. Dose level 4: 2.5 mg daily for days 1-7, 15 mg daily for days 8-21
  Other Names: Revlimid

SUMMARY:
Phase I Study of Lenalidomide in Acute Leukemias and Chronic Lymphocytic Leukemia.

DETAILED DESCRIPTION:
Rationale:

Lenalidomide has properties of thalidomide and appears to have some activity against cancer in laboratory tests. Researchers are still learning how lenalidomide works against cancer in patients. Some ways that this drug seems to produce anti-cancer effects include through stimulating the immune system and blocking blood vessels contributing to cancer growth. The current study will explore different dose levels in patients to gather more information about lenalidomide.

Purpose:

This study will assess the maximum tolerated dose of lenalidomide in patients with relapsed or refractory acute leukemias and chronic lymphocytic leukemias. Toxicity or side effects within patients will also be evaluated. Other purposes of this study include analyzing preliminary clinical activity, pharmacokinetics, and pharmacodynamics. Pharmacokinetics refers to the activity of drugs in the body over a period of time, including how drugs are absorbed, distributed, localized in tissues, and excreted. Pharmacodynamics refers to the bodily processes that lead the drug to effect cancer and other cellular components in the body.

Treatment:

Study participants will be given lenalidomide through intravenous infusions once every 28 days. A 28-day period constitutes a cycle. Since this study will assess the maximum tolerated dose of lenalidomide, some study participants will receive different amounts of this drug compared to others depending upon when each individual enrolls in the study. Each group of 3 to 6 study participants will receive a higher dose of lenalidomide until the maximum tolerated dose is established. Several tests will be performed throughout the study, including bone marrow biopsies. Imaging exams will be conducted as well. Treatments will be discontinued due to disease growth or intolerable adverse effects. Lenalidomide administration will be repeated for 12 or more cycles in patients that experience clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Blood blast count must be < 40,000/uL prior to initiation of therapy. Hydroxyurea (up to 6g/day) may be administered prior to initiation of therapy and during the first week to maintain blood blast count < 40,000/uL
* ECOG(Eastern Cooperative Oncology Group)performance status 0-2.
* Patients with CNS(central nervous system)involvement will be considered eligible for this study if no residual leukemic cells are detected in the CSF (cerebrospinal fluid)following intrathecal chemotherapy or radiation.

Exclusion Criteria:

* Patients with acute promyelocytic leukemia are excluded unless patient has failed salvage therapy with arsenic.
* Patients with HIV are excluded due to increased risk of infectious complications, marrow suppression, and potential interactions with antiviral therapy.
* CLL patients who have had chemotherapy (with the exception of hydroxyurea) or radiotherapy within 4 weeks prior to entering the study are excluded. CLL patients receiving corticosteroids (within 2 weeks) for treatment of disease (other than autoimmune manifestations of CLL) are not eligible.
* Patients who have received mitomycin C or nitrosourea require a six weeks recovery period before they can be enrolled on the current study.
* Patients with the following abnormal clinical values are excluded (unless abnormalities in these parameters are directly attributable to malignancy): Serum creatinine >2.0 mg/dl Total bilirubin > 2 x upper limit of normal (unless due to Gilbert's syndrome) ALT and AST > 5 x upper limit of normal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2007-04 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Maximum tolerable dose | Every 2 weeks during cycle 1; Monthly during subsequent cycles
Toxicities of lenalidomide | Every 2 weeks during cycle 1; Monthly for subsequent cycles

SECONDARY OUTCOMES:
preliminary clinical activity | Twice weekly during cycle 1; Weekly during cycles 2-6; Monthly thereafter
plasma and cellular pharmacokinetics | Days 1, 8, 15 and 21 of first cycle.
pharmacodynamics | Days 1, 8 and 26.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Andritsos, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Result] Maddocks K, Ruppert AS, Browning R, Jones J, Flynn J, Kefauver C, Gao Y, Jiang Y, Rozewski DM, Poi M, Phelps MA, Harper E, Johnson AJ, Byrd JC, Andritsos LA. A dose escalation feasibility study of lenalidomide for treatment of symptomatic, relapsed chronic lymphocytic leukemia. Leuk Res. 2014 Sep;38(9):1025-9. doi: 10.1016/j.leukres.2014.05.011. Epub 2014 May 29. PMID 25082342
- [Derived] Lapalombella R, Andritsos L, Liu Q, May SE, Browning R, Pham LV, Blum KA, Blum W, Ramanunni A, Raymond CA, Smith LL, Lehman A, Mo X, Jarjoura D, Chen CS, Ford R Jr, Rader C, Muthusamy N, Johnson AJ, Byrd JC. Lenalidomide treatment promotes CD154 expression on CLL cells and enhances production of antibodies by normal B cells through a PI3-kinase-dependent pathway. Blood. 2010 Apr 1;115(13):2619-29. doi: 10.1182/blood-2009-09-242438. Epub 2009 Nov 24. PMID 19965642
- [Derived] Fehniger TA, Byrd JC, Marcucci G, Abboud CN, Kefauver C, Payton JE, Vij R, Blum W. Single-agent lenalidomide induces complete remission of acute myeloid leukemia in patients with isolated trisomy 13. Blood. 2009 Jan 29;113(5):1002-5. doi: 10.1182/blood-2008-04-152678. Epub 2008 Sep 29. PMID 18824593
- See also: Jamesline — http://cancer.osu.edu